CLINICAL TRIAL: NCT02956980
Title: Impact of Gender and Pubertal Status on Human Plasmacytoid Dendritic Cells - PLASMACYTOKID Study
Brief Title: Impact of Gender and Pubertal Status on Human Plasmacytoid Dendritic Cells. PLASMACYTOKID
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment target not obtained
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: RC31/16/8251; AOL 2016 (Other Grant/Funding Number: University Hospital Toulouse)
Record Dates: First submitted 2016-11-03; First posted 2016-11-07 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Innate Immune Responses
Keywords: type 1 interferons; children; gender; pubertal status; sex difference
MeSH Terms: conditions — Coitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: non-pubescent children (Experimental): 70 non-pubescent children (25 healthy boys, 25 healthy girls, 10 boys with Klinefelter syndrome and 10 girls with Turner syndrome) Two 7 ml tubes of blood will be taken to perform the functional assays as well as the quantification of Blood Plasmacytoid dendritic cells (pDCs) absolute number in this 70 non-pubescent children.
  Interventions: Biological: Blood Plasmacytoid dendritic cells (pDCs) absolute number
- Group 2: pubescent healthy children (Experimental): 50 pubescent healthy children (25 boys and 25 girls) Two 7 ml tubes of blood will be taken to perform the functional assays as well as the quantification of Blood Plasmacytoid dendritic cells (pDCs) absolute number in this 50 pubescent healthy children.
  Interventions: Biological: Blood Plasmacytoid dendritic cells (pDCs) absolute number

INTERVENTIONS:
Biological: Blood Plasmacytoid dendritic cells (pDCs) absolute number — Two 7 ml tubes will be necessary to perform the functional assays as well as the quantification of blood pDCs absolute number. Functional assays will be performed on isolated PBMC by Ficoll procedure. Quantification of blood pDCs absolute number will be performed on whole blood. After written parental consent, blood sample will be performed on children participating to the study.

SUMMARY:
Differences in pDCs function related to gender have been demonstrated in adults but have never been addressed in children. Yet, differences in immune responses related to gender also exist in children, both in responses to pathogens and susceptibility to autoimmune diseases. The investigators suppose that these differences are partly linked to difference in pDCs functions. This study aim is to compare pDCs functions in children based on gender and pubertal status. This study will be performed in healthy children, boys with Klinefelter syndrome and girls with Turner syndrome.

DETAILED DESCRIPTION:
There are differences in immune responses according to gender. Women have stronger responses against pathogens, especially viruses but are also more susceptible to develop autoimmune diseases. These points reflect more robust innate and adaptive responses in women. Plasmacytoid dendritic cells (pDCs) are key actor of innate immune responses through their ability to produce large amounts of type 1 Interferons (IFN1) secondary to stimulation of their toll like receptors (TLR) 7 and 9 by nucleic acids. Thus, pDCs play a major beneficial role in antiviral responses. In autoimmune diseases like Systemic Erythematous Lupus, pDCs also play a role, mostly deleterious, through inappropriate production of IFN1 upon stimulation of their TLR's by self nucleic acids. In these diseases, pDCs from women have been demonstrated to produce more IFN1 as compared to men, a phenomenon that can be linked to both hormonal and genetic factors. Indeed, the investigators research team demonstrated that IFN1 production by human pDCs can be increased by oestradiol through a specific receptor present in pDCs. Regarding genetics, some studies recently shown in a humanized mouse model, that pDCs developing from female hematopoietic precursor cells have an enhanced TLR 7 mediated IFN1 response as compared to male ones. These results indicate that X chromosome dosage could contribute independently to the enhanced TLR 7 mediated response of pDCs from women. Although some genes implicated in IFN1 production are on the X chromosome, including TLR 7, the mechanism underlying this observation are presently unknown.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patients (0-18 years old):

   * Group 1 : Age<8 years old
   * Group 2 : Age>12 years old
2. Body weight >10kgs
3. Pubescent (group 2) or non-pubescent (group 1)
4. Written consent of parents

Exclusion Criteria:

1. Active infectious disease
2. Known perturbations of immune and/or inflammatory systems
3. Oral or subcutaneous contraception in pubescent girls

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 78 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
percentage of IFN1 producing pDCs | 1 day
  Assessment of the percentage of IFN1 producing pDCs after ex vivo stimulation with TLR 7, 9 and 8 ligands.

SECONDARY OUTCOMES:
Percentage of IFN1 producing tumor necrosis factor(TNF)-alpha | 1 day
  Innate immune functions of pDCs present in the circulating blood of healthy children will be assessed by the percentage of pDCs producing TNF-alpha.
IFN1 concentration in the peripheral blood mononuclear cells circulating (PBMC) culture supernatant. | 1 day
  The innate immune functions of pDCs present in the circulating blood of healthy children will also be assessed by measuring the concentration IFN1 present in the culture supernatant of PBMC stimulated with TLR 7 or TLR 9 ligands.
percentage of cells producing TNF alpha and Interleukin(IL)-12p40 | 1 day
  Innate immune functions of conventional dendritic cells (cDC) and monocytes present in the circulating blood of healthy children will be assessed by the percentage of cells producing TNF alpha and IL-12p40.
percentage of pDc, cDC and monocytes in circulating blood | 1 day
  Innate immune functions of pDCs, cDC and Monocytes present in the circulating blood of boys with Klinefelter syndrome or girls with Turner syndrome will be evaluated identically to healthy children.
Number of DC (cDC and pDC) by milliliter of blood | 1 day
  The number of DCs (pDCs CDC) / ml of blood flowing will be quantified and expressed in blood and percentage of PBMCs.

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Garnier, MD, Principal Investigator — CHU Toulouse, Hôpital des Enfants
Locations (1):
- CHU Toulouse, Hôpital des Enfants, Toulouse, France

IPD SHARING:
Plan to Share IPD: No